CLINICAL TRIAL: NCT03639246
Title: A Phase 1b/2 Randomized, Controlled Study of AVB-S6-500 in Combination With Pegylated Liposomal Doxorubicin (PLD) or Paclitaxel (Pac) in Patients With Platinum-resistant Recurrent Ovarian Cancer
Brief Title: Efficacy and Safety Study of AVB-S6-500 in Patients With Platinum-Resistant Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aravive, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVB500-OC-002
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; Platinum resistant
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel; Chromosomes, Artificial, P1 Bacteriophage; liposomal doxorubicin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 1b: AVB-S6-500+PLD (Experimental)
  Interventions: Drug: AVB-S6-500; Drug: Pegylated liposomal doxorubicin (PLD)
- Phase 1b: AVB-S6-500+Pac (Experimental)
  Interventions: Drug: AVB-S6-500; Drug: Paclitaxel (Pac)
- Phase 2: AVB-S6-500+PLD (Experimental)
  Interventions: Drug: AVB-S6-500; Drug: Pegylated liposomal doxorubicin (PLD)
- Phase 2: AVB-S6-500+Pac (Experimental)
  Interventions: Drug: AVB-S6-500; Drug: Paclitaxel (Pac)
- Phase 2: Placebo+PLD (Active Comparator)
  Interventions: Drug: Pegylated liposomal doxorubicin (PLD); Other: Placebo
- Phase 2: Placebo+Pac (Active Comparator)
  Interventions: Drug: Paclitaxel (Pac); Other: Placebo

INTERVENTIONS:
Drug: AVB-S6-500 — AVB-S6-500 is experimental drug
  Arms: Phase 1b: AVB-S6-500+PLD; Phase 1b: AVB-S6-500+Pac; Phase 2: AVB-S6-500+PLD; Phase 2: AVB-S6-500+Pac
Drug: Paclitaxel (Pac) — Paclitaxel is active comparator
  Other Names: Taxol
  Arms: Phase 1b: AVB-S6-500+Pac; Phase 2: AVB-S6-500+Pac; Phase 2: Placebo+Pac
Drug: Pegylated liposomal doxorubicin (PLD) — PLD is active comparator
  Other Names: Doxil
  Arms: Phase 1b: AVB-S6-500+PLD; Phase 2: AVB-S6-500+PLD; Phase 2: Placebo+PLD
Other: Placebo — Placebo comparator
  Arms: Phase 2: Placebo+PLD; Phase 2: Placebo+Pac

SUMMARY:
This is a Phase 1b/2 study of AVB-S6-500 in combination with pegylated liposomal doxorubicin (PLD) or paclitaxel (Pac) in patients with platinum resistant recurrent ovarian cancer. The phase 1b portion of the study is open label and patients will receive either AVB-S6-500+PLD or AVB-S6-500+ Pac. The Phase 2 portion of the study is randomized, double-blind, placebo-controlled study to compare efficacy and tolerability of AVB-S6-500 in combination with PLD or Pac versus placebo plus PLD or Pac.

DETAILED DESCRIPTION:
While this study was planned as two-part study consisting of a Phase 1b and a Phase 2 portion, the sponsor decided not to proceed with the Phase 2 portion.

The Phase 1b portion of the study was a multicenter, 2-group, open-label design to evaluate the safety and tolerability of AVB-S6-500 combined with PLD or Pac in subjects with platinum-resistant recurrent ovarian cancer. The decision to enroll in the Phase 2 portion of the study was to be driven by the recommendation of a safe and tolerable dose of AVB-S6-500 in combination with each chemotherapy backbone; however, enrollment into the Phase 2 portion was not initiated per Sponsor decision. Given that sufficient data were obtained in the Phase 1b portion AVB-S6-500 + Pac group, the decision was made to pursue a randomized Phase 3 to further study the benefit of this combination versus paclitaxel alone in patients with platinum resistant ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Histologically confirmed and documented recurrent ovarian, fallopian tube, and peritoneal cancer.
* Platinum resistant disease, defined as progression within ≤ 6 months from completion of most recent regimen and calculated from the date of the last administered dose of platinum therapy
* Must have available archived tumor tissue OR if archived tissue is not available, willing to provide a fresh tumor biopsy
* Must have radiologic imaging with a computerized tomography (CT) scan or magnetic resonance imaging (MRI) within 4 weeks of first dose of study drug
* Received at least 1 but not more than 3 therapy regimens, not including maintenance or adjuvant therapy
* Must have ovarian cancer that is measurable according to RECIST 1.1
* ECOG performance status of 0-1
* Normal gastrointestinal (GI), bone marrow, liver and kidney function
* At least 28 days between termination of prior anti-cancer or hormonal therapy and administration of AVB-S6-500

Exclusion Criteria:

* Primary platinum-refractory disease (defined as progression during the first platinum regimen or within 4 weeks of completion of the first platinum regimen)
* Currently being treated with concurrent anti-cancer therapy or any other interventional treatment or trial
* Received prior therapy with Pac or PLD in the recurrent setting, depending on physician-chosen chemotherapy for this study
* Significant cardiac disease history
* Has other prior or concurrent malignancy within the past 5 years except adequately treated basal cell skin cancer or carcinoma in situ of the cervix
* Symptomatic CNS metastasis or metastases
* Serious active infection requiring IV antibiotics and/or hospitalization at study entry
* Has known previous or current human immune deficiency (HIV) syndrome, hepatitis B, or hepatitis C
* Has had paracentesis for ascites within 3 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | 6 months
  Measured by the number of patients with AEs in Phase 1 portion of the study.
Anti-tumor activity of AVB-S6-500 in combination with PLD | 18 months
  Measured by progression free survival (PFS) in patients receiving AVB-S6-500+PLD versus patients receiving Placebo+PLD in Phase 2 portion of the study.
Anti-tumor activity of AVB-S6-500 in combination with Pac | 18 months
  Measured by progression free survival (PFS) in patients receiving AVB-S6-500+ Pac versus patients receiving Placebo+Pac in Phase 2 portion of the study.

SECONDARY OUTCOMES:
Pharmacokinetics: AUC | 18 months
  Area under the AVB-S6-500 concentration-time curve.
Pharmacokinetics: Cmax | 18 months
  Maximum observed AVB-S6-500 concentration.
Pharmacokinetics: Tmax | 18 months
  Time of maximum observed AVB-S6-500 concentration.
Pharmacokinetics: t1/2 | 18 months
  Apparent terminal half-life of AVB-S6-500.
Pharmacodynamic marker assessment | 18 months
  Change from the baseline in GAS6 serum levels.
Anti-drug antibody (ADA) titers | 18 months
  Change from baseline in ADA titer.
Objective response rate | 18 months
  Proportion of subjects who have a partial or complete response to therapy relative to baseline as assessed per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as well as Gynecologic Cancer Intergroup (GCIG) cancer antigen (CA)-125 criteria.
Disease control rate | 18 months
  Proportion of subjects who have a complete or partial response to therapy or maintain stable disease.
Duration of response (DOR) | 18 months
  Measured from the date of partial or complete response to therapy until the cancer progresses.
Overall survival | 30 months
  Time following the treatment until death.
CA-125 response rate | 18 months
  Proportion of subjects with a minimum 50% reduction in CA-125 serum levels lasting for 28 days relative to baseline CA-125 serum levels.
Quality of Life(QOL) | 18 months
  Subject QOL will be assessed every 8 weeks during treatment using the Functional Assessment Of Cancer Therapy - Ovarian Cancer (FACT-O) questionnaire, which consists of 4 subscales: physical well-being (7 questions), social/family well-being (7 questions), emotional well-being (6 questions), and functional well-being (7 questions), and 12 additional concerns specific to ovarian cancer. All items are rated on a 5 point scale with 0 "not at all" and 4 "very much". The scoring algorithm allows for eight summary scales: the four core well-being subscales, a subtotal of the 27 core items, a subtotal of the 12 ovarian-specific additional concerns, a grand total of the 39 items, and a trial outcome index (sum of the 17 physical and functional wellbeing items plus the 12 ovarian-specific items).

CONTACTS AND LOCATIONS:
Overall Officials: Amy Franke, Study Director — Aravive, Inc.
Locations (16):
- United States (16):
  - Arizona Oncology, Phoenix, Arizona
  - Arizona Oncology Associates, Tucson, Arizona
  - Kaiser Permanente Oakland, Oakland, California
  - Kaiser Permanente Roseville, Roseville, California
  - Kaiser Permanente San Francisco, San Francisco, California
  - Kaiser Permanente Santa Clara, Santa Clara, California
  - Kaiser Permanente Vallejo, Vallejo, California
  - Kaiser Permanente Walnut Creek, Walnut Creek, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - OUHSC-Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Texas Oncology - Austin Central, Austin, Texas
  - Texas Oncology - Fort Worth, Fort Worth, Texas
  - Texas Oncology - San Antonio Medical Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No